CLINICAL TRIAL: NCT06162533
Title: SARS-CoV-2 Re-Infection Risk and Vaccine Efficacy in Austria: SARIVA Study
Brief Title: Severe Acute Respiratory Syndrome Coronavirus 2 Re-Infection Risk and Vaccine Efficacy in Austria
Acronym: SARIVA
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: AGES (Unknown); Medical University Innsbruck (Other); Austrian Science Fund (FWF) (Other)
Responsible Party: Sponsor
Other Study IDs: SARIVA 1.0.
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Vaccinated against SARS-CoV-2: Individuals who received a SARS-CoV-2 vaccine but have no record of a previous SARS-CoV-2 infection.
  Subgroups will be formed according to the number and type of vaccines against SARS-CoV-2.
  Interventions: Biological: Vaccination against SARS-CoV-2
- Previously SARS-CoV-2 infected: Individuals who were previously infected with SARS-CoV-2 but have not received a SARS-CoV-2 vaccine.
  Subgroups will be formed according to the number and time period of previous SARS-CoV-2 infections.
- Hybrid Immunity against SARS-CoV-2: Individuals who received a SARS-CoV-2 vaccine and who were previously infected with SARS-CoV-2.
  Subgroups will be formed according to the number and time period of previous SARS-CoV-2 infections, the number and type of vaccines against SARS-CoV-2, and according to whether the vaccination or the infection was the first immune conferring event.
  Interventions: Biological: Vaccination against SARS-CoV-2
- No immunity against SARS-CoV-2: Individuals who have not received a SARS-CoV-2 vaccine and were not previously infected with SARS-CoV-2.

INTERVENTIONS:
Biological: Vaccination against SARS-CoV-2 — Interventions are either a vaccination against SARS-CoV-2 or an infection with SARS-CoV-2
  Other Names: Infection with SARS-CoV-2
  Groups: Hybrid Immunity against SARS-CoV-2; Vaccinated against SARS-CoV-2

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic was caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) virus. In this study, we aim to evaluate how strong and how long are individuals in Austria after vaccination and/or infection with SARS-CoV-2 protected against COVID-19 disease.

In this project, we will analyze national health data from all inhabitants of Austria (about 9 million persons) during the COVID-19 pandemic. The population of Austria will be stratified into different groups according to previous vaccinations against SARS-CoV-2 and previous SARS-CoV-2 infections.

We primarily evaluate how strong and how long after vaccination against SARS-CoV-2 and/or infection with SARS-CoV-2, the risk for COVID-19 deaths is reduced or altered as compared to less vaccinated and/or infected persons. As secondary study aims, we perform such analyses also for SARS-CoV-2 infections, hospitalizations and intensive care unit (ICU) stays, with or due to SARS-CoV-2. These analyses will be performed during different time periods of the COVID-19 pandemic, and we will also perform various subgroup analyses as for example according to age and gender. Given that antibodies against SARS-CoV-2 are usually detected after vaccination and/or infection, we will use such antibody data from blood donors in Tyrol, to elucidate how well the national health data on SARS-CoV-2 infections and vaccinations match with the respective antibody data, and how well these antibody data indicate risk of COVID-19 deaths and infections.

We will calculate the probability of dying due to a SARS-CoV-2 infection (case/infection fatality rate) for different times of the COVID-19 pandemic, in order to document the health threat due to SARS-CoV-2. Based on all these data, we will calculate how many persons have to be vaccinated against SARS-CoV-2 to prevent one COVID-19 death at different times during this COVID-19 pandemic. We will consider the respective COVID-19 policies such as mask mandates, lock-downs, SARS-CoV-2 test mandates in our analyses and will evaluate the impact of these policies on COVID-19 deaths and diseases. In addition, we will evaluate data on total mortality according to the number of SARS-CoV-2 vaccinations and/or infections, and we will aim to collaborate with other research groups in order to extend our analyses.

In conclusion, the results of this study should provide an overview on the COVID-19 pandemic with respect to protection conferred by vaccinations and previous SARS-CoV-2 infections, as well as the health threat of SARS-CoV-2, in order to provide knowledge for future COVID-19 policy and future pandemics.

ELIGIBILITY:
Inclusion Criteria:

- Residency in Austria.

Exclusion Criteria:

- None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The national population of Austria
Sampling Method: Probability Sample
Enrollment: 9090868 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
COVID-19 death | January 1, 2000 to June 30, 2023
  Death due to COVID-19

SECONDARY OUTCOMES:
SARS-CoV-2 infection | January 1, 2000 to June 30, 2023
  Documented SARS-CoV-2 infection
ICU stay | January 1, 2000 to June 30, 2023
  ICU stay of COVID-19 patients
Hospitalization | January 1, 2000 to June 30, 2023
  Hospitalization of COVID-19 patients
All-cause mortality | January 1, 2000 to June 30, 2023
  Death due to all-causes

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Austrian Agency for Health and Food Safety, Vienna

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data of this study are available upon request with approval needed from the Austrian Agency for Health and Food Safety (AGES), Vienna, Austria, and an ethical approval or waiver by the local ethic committee for use of these data. The individual participant data are not publicly available due to restrictions pertaining to contained information that could compromise the privacy of individuals (i.e. potentially allow the identification of certain individuals based on e.g. birthdate, gender and infection or death date). Data are stored at the AGES. The same data availability rules apply to the antibody data (i.e. Anti-SARS-CoV-2 antibodies) from the Medical University of Innsbruck.